CLINICAL TRIAL: NCT02863718
Title: A Placebo-Controlled, Double-Blind, Randomized, Multicenter, Three Arm Phase III Trial to Compare the Efficacy and Safety of Ibrutinib Vs. Placebo in Previously Untreated Binet Stage a Chronic Lymphocytic Leukemia Patients with Risk of Early Disease Progression
Brief Title: Ibrutinib in Previously Untreated Binet Stage a Chronic Lymphocytic Leukemia with Risk of Disease Progression
Acronym: CLL12
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLL12; 2013-003211-22 (EudraCT Number)
Record Dates: First submitted 2014-06-10; First posted 2016-08-11 (Estimated); Last update posted 2024-12-30 (Actual); Status verified 2022-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Watch & wait (No Intervention): Watch & wait
- Placebo 420 mg/d (Placebo Comparator): Placebo 420mg/d
  Interventions: Drug: Placebo
- Ibrutinib 420mg/d (Active Comparator): Ibrutinib 420mg/d
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Bruton's tyrosine kinase Inhibitor Ibrutinib 420mg daily
  Other Names: Imbruvica
  Arms: Ibrutinib 420mg/d
Drug: Placebo — Placebo 420mg daily
  Arms: Placebo 420 mg/d

SUMMARY:
This is a prospective, multicenter, randomized, placebo-controlled, double-blind phase III study that compares the efficacy and safety of oral ibrutinib in previously untreated Binet stage A CLL patients without treatment indication according to iwCLL guidelines but risk of early disease progression.

For event-free survival (EFS), an improvement from 24 months for untreated intermediate or (very) high risk CLL to 48 months for subjects treated with ibrutinib is considered clinically relevant. Ibrutinib / placebo is administered continuously orally until symptomatic disease progression, unacceptable toxicity, or voluntary treatment withdrawal, whichever occurs first.

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate superiority of ibrutinib over placebo in prolonging EFS for subjects with treatment-naïve CLL stage A and intermediate or (very) high risk of disease progression. All subjects with intermediate, (very) high risk randomized to the experimental treatment arm will be treated up to active progressive disease with treatment indication according to iwCLL-Guidelines with the objective to demonstrate prolongation of EFS for the ibrutinib arm. EFS is defined as the time between randomization until active progressive disease with treatment indication according to the iwCLL-Guidelines with subsequent treatment for CLL or death.

The secondary objectives are:

* To evaluate the prolongation of overall survival of ibrutinib versus placebo
* To evaluate the safety of ibrutinib versus placebo

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated CLL
* Stage Binet A without need for treatment
* Age ≥ 18 years
* Life expectancy ≥ 6 months
* ECOG 0 - 2
* Signed written informed consent
* Patient in the experimental arm is willing to use a highly effective contraceptive method
* Male subjects in the experimental treatment arm (placebo / ibrutinib) must:
* Agree to not donate semen during study drug therapy and for a period after end of study drug therapy.
* For males these restrictions apply for 3 months after the last dose of study medication.
* Agree not to share study medication with another person.
* Be counseled about pregnancy precautions and risks of fetal exposure.
* Willingness to inform the general practitioner

Exclusion Criteria:

* Any prior CLL specific therapy
* Prior treatment with Ibrutinib or BTK inhibitors
* Chronic use of steroids in excess of prednisone 20mg/day or its equivalent
* Active infections requiring systemic antibiotics
* An life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion could compromise the subject's safety, interfere with the absorption or metabolism of Ibrutinib capsules, or put the study outcomes at undue risk
* Pregnant or lactating females
* Central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging. Subjects who have signs or symptoms suggestive of leukemic meningitis or a history of leukemic meningitis must have a lumbar puncture procedure performed within two weeks prior to randomization
* Known second malignancy that limits survival to less than two years
* Known Human Immunodeficiency Virus (HIV), active Hepatitis B Virus (HBV) and/or active Hepatitis C Virus (HCV) infection.
* Any of the following laboratory abnormalities:

  1. Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 2.5 x upper limit of normal (ULN)
  2. Serum total bilirubin > 1.5 ULN (with the exception of Gilbert's Syndrome)
  3. Creatinine clearance < 30ml/min
* Requires anticoagulant with warfarin or phenoprocoumon
* Requires anticoagulant with oral direct Xa Inhibitors (rivaroxaban, apixaban, edoxaban)
* History of stroke or intracranial hemorrhage within 6 months prior to randomization
* Requires treatment with strong CYP3A4/5 Inhibitors
* Participation in any clinical study for CLL or having taken any investigational therapy which would interfere with the study drug for a disease other than CLL within 28 days prior to initiating treatment.
* Prisoners or subjects who are institutionalized by regulatory or court order or persons who are in dependence to the sponsor or an investigator
* Patients with uncontrolled autoimmune hemolytic anemia or autoimmune thrombocytopenia
* For males these restrictions apply for 3 months after the last dose of study medication.
* Agree not to share study medication with another person.
* Be counseled about pregnancy precautions and risks of fetal exposure.
* Willingness to inform the general practitioner
* Requires anticoagulant with warfarin or phenoprocoumon
* Requires anticoagulant with oral direct Xa inhibitors (rivaroxaban, apixaban, edoxaban)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2014-04-30 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2022-07-11 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | randomization until progression, initiation of subsequent treatment for CLL or death by any cause, whichever occurs first, assessed for at at least 60 months
  EFS is defined as the time between the date of completed registration and time point of symptomatic disease progression with treatment indication, initiation of subsequent treatment for CLL or death by any cause, whichever occurs first. These will be counted as event for EFS.

SECONDARY OUTCOMES:
Treatment-free survival | time of randomization until the date of initiation of subsequent treatment for CLL or death by any cause assessed for at at least 60 months
  The primary efficacy parameter is event-free survival (EFS) defined as the time of randomization until symptomatic disease progression with treatment indication, initiation of subsequent treatment for CLL or death by any cause, whichever occurs first
Progression-free survival (PFS) | the time of randomization until symptomatic disease progression (as defined by the updated iwCLL-guidelines) or death by any cause, whichever occurs first, assessed for at at least 60 months
  PFS is defined by the time of randomization until symptomatic disease progression (as defined by the updated iwCLL-guidelines) or death by any cause, whichever occurs first. These will be counted as event for PFS. Patients for whom no documented event for PFS is available at the time of analysis will be censored at the time point of last follow-up information they were assessed to be event-free.
Response rates (Overall response rate (ORR); Complete Remission (CR); Partial Remission (PR) | Overall response rate (ORR) achieved during treatment or within 6 months of end of treatment, complete response (CR) and partial response (PR) rates will be evaluated for at least 60 months or Progression whichever occurs first
  ORR, CR- and PR- rates are defined by the proportion of patients having achieved a response (CR/CRi and nPR/PR), CR/CRi and nPR/PR as best response respectively based on the respective population.
rate of Treatment-related adverse events | randomization until 28 days after the last dose of study drug
Overall survival (OS) | date of randomization to the date of death for at least 60 months
  Respectively, for watch & wait- patients (study arm I) the date of completed registration will be used. Additionally, OS will also be calculated for the time period between first diagnosis of CLL and death due to any cause. Subjects who have not yet died at the time of analysis will be censored at the time of last follow-up information they were assessed to be alive.
  The exact cause of death will be recorded, with additional differentiation between CLL-related, treatment-related and other causes.
  Furthermore overall survival will be analyzed using a multivariate Cox regression model adjusted for risk category, study arm, and baseline prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Petra Langerbeins, MD, Principal Investigator — German CLL Study Group
Locations (1):
- German CLL Study Group, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langerbeins P, Robrecht S, Nieper P, Cramer P, Furstenau M, Al-Sawaf O, Simon F, Fink AM, Kreuzer KA, Vehling-Kaiser U, Tausch E, Schneider C, Muller L, Eckart MJ, Schlag R, Freier W, Gaska T, Balser C, Reiser M, Stauch M, Zahn MO, Dorfel S, Staib P, Behlendorf T, Hensel M, Hebart H, Klaproth H, Block A, Liersch R, Hauch U, Heinrich B, Wendtner CM, Fischer K, Stilgenbauer S, Eichhorst B, Hallek M. Ibrutinib in Early-Stage Chronic Lymphocytic Leukemia: The Randomized, Placebo-Controlled, Double-Blind, Phase III CLL12 Trial. J Clin Oncol. 2025 Feb;43(4):392-402. doi: 10.1200/JCO.24.00975. Epub 2024 Nov 27. PMID 39602678
- [Background] Langerbeins P, Zhang C, Robrecht S, Cramer P, Furstenau M, Al-Sawaf O, von Tresckow J, Fink AM, Kreuzer KA, Vehling-Kaiser U, Tausch E, Muller L, Eckart MJ, Schlag R, Freier W, Gaska T, Balser C, Reiser M, Stauch M, Wendtner CM, Fischer K, Stilgenbauer S, Eichhorst B, Hallek M. The CLL12 trial: ibrutinib vs placebo in treatment-naive, early-stage chronic lymphocytic leukemia. Blood. 2022 Jan 13;139(2):177-187. doi: 10.1182/blood.2021010845. PMID 34758069